CLINICAL TRIAL: NCT01680328
Title: Investigation of Pain During Subcutaneous Injections With Different Injection Speed and Volume Combinations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: INS-4011; U1111-1129-4191 (Other: WHO)
Record Dates: First submitted 2012-08-31; First posted 2012-09-07 (Estimated); Results first posted 2014-06-19 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Sodium Chloride; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Different injection speed and volume combinations (Other): The study consists of 80 treatment arms in a cross-over design with 19 treatments and 19 periods. The 80 treatment arms will represent different orders of the 19 treatments and each treatment arm will be used for one subject. A subject not completing all treatments will be replaced by another subject using the same treatment arm.
  Interventions: Other: 19 injections; Drug: sodium chloride 0.9% solution

INTERVENTIONS:
Other: 19 injections — Subjects will receive 19 injections in randomised order of which 13 will be in the abdomen and 6 in the thighs. Out of the 19 injections, 2 are needle insertions only. The remaining 17 injections represent different combinations of injection speed and volume of sodium chloride 0.9% solution for injection. The order of the injection speed and volume combinations will be blinded for the subject and the pain will be evaluated by the subject on a VAS (Visual Analogue Scale).
Drug: sodium chloride 0.9% solution — Solution for injection.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to assess and describe the pain in relation to subcutaneous (under the skin) injection of different combinations of injection speed and volume with respect to acceptance of the injection pain and backflow.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities.
* Type 1 or type 2 diabetes
* Daily injection(s) with anti-diabetic drug (insulin or Glucagon like Peptide-1 (GLP-1) analogues) via pen-injector or vial/syringe for more than 6 months
* Body mass index (BMI) between 18.5 and 30.0 kg/m^2 (both included)
* Caucasians

Exclusion Criteria:

* Known or suspected hypersensitivity to needle, ink ball pen or other that are in contact with the injection area during the clinical visit
* Previous participation in this trial. Participation is defined as: screened
* Receipt of any investigational medicinal product that can influence pain perception within 14 days before screening
* Injection of more than 40 units of insulin per injection
* Continuous Subcutaneous Insulin Infusion use within the last 6 months
* Continuous Glucose Monitoring use within the last 6 months
* Intake of any pain-relieving or analgesic within the last week (excluding low dose aspirin in cardio vascular prophylactic doses)
* Known active or in-active skin disease in the injection area or that may affect pain perception
* Anti-coagulant treatment within the last month (low dose of aspirin in cardiovascular prophylactic doses is allowed. However, not on the day of the injections)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Nosek L, Dellweg S, Zijlstra E, Praestmark KA, Kildegaard J, Nielsen G, Sparre T. Impact of injection speed and volume on perceived pain during subcutaneous injections into the abdomen and thigh: a single-centre, randomized controlled trial. Diabetes Obes Metab. 2014 Oct;16(10):971-6. doi: 10.1111/dom.12304. Epub 2014 May 11. PMID 24720741
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at a single site in Germany at a single visit.
Groups:
- All Participants: Subjects received 19 subcutaneous (s.c) injections. Of the 19 injections, 13 were in the abdomen and 6 in the thighs. Of the 13 injections in the abdomen, 1 was a needle insertion and 12 were combinations of the 4 different injection volumes (400, 800, 1200 and 1600 µL) and 3 injection speeds (150, 300 and 450 µL/s). Of the 6 injections in the thigh, 1 was a needle insertion and 5 were selected combinations of injection volume (µL) and speed (µL/s) (400/150, 400/450, 800/300, 1600/150, 1600/450). Except for the 2 needle insertions, sodium chloride 0.9% solution was injected.
Period: Overall Study
Arm/Group | All Participants
Started | 82
Subjects Missing Injections | 2 (One missed the [1600 μL, 450 μL/s; thighs]; one missed the [400 μL, 300 μL/s; abdomen])
Completed | 80
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.9)
Gender [Count of Participants; unit: Participants]
  Female | 32
  Male | 50

OUTCOME MEASURES:

1. Primary Outcome: Injection Pain (VAS mm)
Description: Calculated as the least square mean estimate of the difference in injection pain on a VAS (mm) between different factor levels corresponding to injection region, injection volume and injection speed (pain was assessed using an electronic VAS consisting of a 100 mm line where 0 mm corresponded to no pain and 100 mm corresponded to worst pain. After each injection, the subjects rated their pain perception at the electronic VAS by marking the 100 mm line).
Time Frame: 1 minute (±30 sec) after each injection
Population: All randomised subjects receiving at least one injection (possibly needle insertion only) were included in the full analysis set. A total of 4 subjects did not contribute to the analysis due to missing injections (2) and missing VAS evaluation (2).
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Thighs: Injection Region-5 s.c Injections+1 Needle Insertion: Pain (VAS) was assessed in each subject for the 5 s.c injections+1 needle insertion administered in the thighs.
- Abdomen: Injection Region-12 s.c Injections+1 Needle Insertion: Pain (VAS) was assessed in each subject for the 12 s.c injections+1 needle insertion administered in the abdomen.
- Injection Volume 1600 μL; Injection Volume 1200 μL; Injection Volume 800 μL; Injection Volume 400 μL; Injection Speed at 450 μL/s; Injection Speed at 300 μL/s; Injection Speed at 150 μL/s: Pain (VAS) was assessed in the abdomen following administration of 4 different injection volumes (400, 800, 1200 and 1600 µL) at 3 different injection speeds (150, 300 and 450 µL/s); and in the thighs following administration of the selected combinations of injection volume (µL) and speed (µL/s) (400/150, 400/450, 800/300, 1600/150, 1600/450).
Arm/Group | Thighs: Injection Region-5 s.c Injections+1 Needle Insertion | Abdomen: Injection Region-12 s.c Injections+1 Needle Insertion | Injection Volume 1600 μL | Injection Volume 1200 μL | Injection Volume 800 μL | Injection Volume 400 μL | Injection Speed at 450 μL/s | Injection Speed at 300 μL/s | Injection Speed at 150 μL/s
Number analyzed (Participants) | 82 | 82 | 82 | 82 | 82 | 82 | 82 | 82 | 82
mm
  Needle insertion | 20.0 (24.2) | 12.8 (16.3) | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered
  Injection speed at 150 μL/s; Abdomen | NA (NA) — Not administered | NA (NA) — Not administered | 20.9 (24.4) | 15.7 (20.2) | 11.6 (15.7) | 14.5 (17.3) | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — No summary statistics done for this combination
  Injection speed at 300 μL/s; Abdomen | NA (NA) — Not administered | NA (NA) — Not administered | 17.2 (22.5) | 20.1 (25.3) | 13.7 (17.1) | 14.8 (18.1) | NA (NA) — Not administered | NA (NA) — No summary statistics done for this combination | NA (NA) — Not administered
  Injection speed at 450 μL/s; Abdomen | NA (NA) — Not administered | NA (NA) — Not administered | 21.1 (24.8) | 14.9 (16.9) | 14.8 (18.9) | 12.4 (15.5) | NA (NA) — No summary statistics done for this combination | NA (NA) — Not administered | NA (NA) — Not administered
  Injection volume of 400 μL; Thighs | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — No summary statistics done for this combination | 20.9 (24.8) | NA (NA) — Not administered | 22.9 (25.9)
  Injection volume of 800 μL; Thighs | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — No summary statistics done for this combination | NA (NA) — Not administered | NA (NA) — Not administered | 23.2 (24.5) | NA (NA) — Not administered
  Injection volume of 1600 μL; Thighs | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — No summary statistics done for this combination | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | 31.1 (28.5) | NA (NA) — Not administered | 31.5 (28.0)
Statistical Analysis 1: Comparison: Injection Volume 800 μL vs Injection Volume 400 μL; Though the sample size was not based on any formal sample size or power calculations as no statistical tests were pre-specified to address the endpoints, a sample size of 80 completers was derived from a simulation study. Mean Difference in injection pain on VAS after injection of different volumes was calculated as least square mean estimate of the mean difference in injection pain; Test type: Superiority or Other; Least Squares Mean = -0.1, 95% CI [-2.9 to 2.8]
Statistical Analysis 2: Comparison: Injection Volume 1200 μL vs Injection Volume 400 μL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Least Squares Mean = 3.5, 95% CI [0.4 to 6.6]
Statistical Analysis 3: Comparison: Injection Volume 1600 μL vs Injection Volume 400 μL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Least Squares Mean = 7.2, 95% CI [4.6 to 9.7]
Statistical Analysis 4: Comparison: Injection Volume 1200 μL vs Injection Volume 800 μL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Least Squares Mean = 3.6, 95% CI [0.4 to 6.7]
Statistical Analysis 5: Comparison: Injection Volume 1600 μL vs Injection Volume 800 μL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Least Squares Mean = 7.2, 95% CI [4.4 to 10.0]
Statistical Analysis 6: Comparison: Injection Volume 1600 μL vs Injection Volume 1200 μL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Least Squares Mean = 3.7, 95% CI [0.6 to 6.7]
Statistical Analysis 7: Comparison: Injection Speed at 300 μL/s vs Injection Speed at 150 μL/s; Though the sample size was not based on any formal sample size or power calculations as no statistical tests were pre-specified to address the endpoints, a sample size of 80 completers was derived from a simulation study. Mean difference in injection pain on VAS after injection at different speeds was calculated as least square mean estimate of the mean difference in injection pain on a VAS after injection at different speeds; Test type: Superiority or Other; Least Squares Mean = 0.4, 95% CI [-2.1 to 2.9]
Statistical Analysis 8: Comparison: Injection Speed at 450 μL/s vs Injection Speed at 150 μL/s; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; Least Squares Mean = -0.4, 95% CI [-2.7 to 1.9]
Statistical Analysis 9: Comparison: Thighs: Injection Region-5 s.c Injections+1 Needle Insertion vs Abdomen: Injection Region-12 s.c Injections+1 Needle Insertion; Though the sample size was not based on any formal sample size or power calculations as no statistical tests were pre-specified to address the endpoints, a sample size of 80 completers was derived from a simulation study. The mean difference in injection pain on a VAS (mm) between the thighs and abdomen was calculated as the least square mean estimate of the mean difference in injection pain on a VAS (mm) between the thighs and abdomen; Test type: Superiority or Other; Least Squares Mean = 9.0, 95% CI [6.7 to 11.3]

2. Secondary Outcome: Acceptance of Injection Pain After Injection of Different Volumes.
Description: Acceptance of pain was rated subjectively as yes or no by the subject after each injection.
Time Frame: 1 minute (±30 seconds) after each injection
Population: All randomised subjects receiving at least one injection (possibly needle insertion only) were included in the full analysis set.
Measure: Number; unit: scores
Groups:
- Injection Volume of 1600 μL; Injection Volume of 1200 μL; Injection Volume of 800 μL; Injection Volume of 400 μL: Acceptance of pain was assessed in each subject for all injections.
Arm/Group | Injection Volume of 1600 μL | Injection Volume of 1200 μL | Injection Volume of 800 μL | Injection Volume of 400 μL
Number analyzed (Participants) | 82 | 82 | 82 | 82
scores
  Yes | 334 | 218 | 303 | 368
  No | 75 | 28 | 25 | 41
Statistical Analysis 1: Comparison: Injection Volume of 800 μL vs Injection Volume of 400 μL; Acceptance of pain was rated subjectively as yes or no by the subject after each injection. The odds are calculated as 'no versus yes', and 'larger volume versus smaller', so that an odds ratio above 1 corresponds to a higher frequency of unacceptable pain for the larger volume - i.e. a worse condition. The odd ratios for unacceptable injection pain are based on a statistical model for all acceptance pain data; Test type: Superiority or Other; Odds ratio (OR); Odds Ratio (OR) = 0.8, 95% CI [0.5 to 1.4]
Statistical Analysis 2: Comparison: Injection Volume of 1200 μL vs Injection Volume of 400 μL; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 2.1, 95% CI [1.2 to 3.5]
Statistical Analysis 3: Comparison: Injection Volume of 1600 μL vs Injection Volume of 400 μL; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 2.1, 95% CI [1.4 to 3.0]
Statistical Analysis 4: Comparison: Injection Volume of 1200 μL vs Injection Volume of 800 μL; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 2.6, 95% CI [1.4 to 4.8]
Statistical Analysis 5: Comparison: Injection Volume of 1600 μL vs Injection Volume of 800 μL; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 2.6, 95% CI [1.4 to 4.6]
Statistical Analysis 6: Comparison: Injection Volume of 1600 μL vs Injection Volume of 1200 μL; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 1.0, 95% CI [0.7 to 1.5]

3. Secondary Outcome: Acceptance of Injection Pain After Injection at Different Speeds.
Description: Acceptance of pain was rated subjectively as yes or no by the subject after each injection.
Time Frame: 1 minute (±30 sec) after each injection
Population: as for outcome 2
Measure: Number; unit: scores
Groups:
- Injection Speed at 450 μL/s; Injection Speed at 300 μL/s; Injection Speed at 150 μL/s: Acceptance of pain was assessed in each subject for all injections.
Arm/Group | Injection Speed at 450 μL/s | Injection Speed at 300 μL/s | Injection Speed at 150 μL/s
Number analyzed (Participants) | 82 | 82 | 82
scores
  Yes | 432 | 365 | 426
  No | 59 | 44 | 66
Statistical Analysis 1: Comparison: Injection Speed at 300 μL/s vs Injection Speed at 150 μL/s; Acceptance of pain was rated subjectively as yes or no by the subject after each injection. The odds are calculated as 'no versus yes', and 'higher speed versus lower', so that an odds ratio above 1 corresponds to a higher frequency of unacceptable pain for the higher speed - i.e. a worse condition. The odd ratios for unacceptable injection pain are based on a statistical model for all acceptance pain data; Test type: Superiority or Other; Odds Ratio (OR) = 1.1, 95% CI [0.7 to 1.8]
Statistical Analysis 2: Comparison: Injection Speed at 450 μL/s vs Injection Speed at 150 μL/s; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.9, 95% CI [0.6 to 1.2]

4. Secondary Outcome: Acceptance of Injection Pain After Injection in the Thighs Versus Abdomen.
Description: Acceptance of pain was rated subjectively as yes or no by the subject after each injection.
Time Frame: 1 minute (±30 seconds) after each injection
Population: as for outcome 2
Measure: Number; unit: scores
Groups:
- Thighs: Acceptance of pain was assessed in each subject for all injections in the thighs.
- Abdomen: Acceptance of pain was assessed in each subject for all injections in the abdomen.
Arm/Group | Thighs | Abdomen
Number analyzed (Participants) | 82 | 82
scores
  Yes | 390 | 978
  No | 101 | 87
Statistical Analysis 1: Comparison: Thighs vs Abdomen; Acceptance of pain was rated subjectively as yes or no by the subject after each injection. The odds are calculated as 'no versus yes', so that an odds ratio above 1 corresponds to a higher frequency of unacceptable pain in the thighs - i.e. a worse condition; Test type: Superiority or Other; Odds ratio (OR); Odds Ratio (OR) = 3.7, 95% CI [2.4 to 5.5]

5. Secondary Outcome: Estimated Mean Differences in the Volume of Backflow (uL) in the Abdomen After Different Injection Volumes and Speeds as Compared to Needle Insertion
Description: Backflow was measured after each injection by placing a filter paper over the injection site after the injection was given and until the liquid was absorbed. The size of the wet spot on the filter paper served as a measure of the backflow. The treatment effect on backflow was calculated as the least square mean estimate of the difference in backflow after injection in the abdomen at different volume and speed combinations.
Time Frame: 2 minutes (±30sec) after each injection
Population: All randomised subjects receiving at least one injection (possibly needle insertion only) were included in the full analysis set. One subject did not contribute to the analysis due to missing injection.
Measure: Mean (Standard Deviation); unit: mcL
Groups:
- Abdomen: Injection Region-12 s.c Injections+1 Needle Insertion: Backflow (uL) was assessed in each subject for the 12 s.c injections+1 needle insertion administered in the abdomen.
- Injection Volume 1600 μL; Injection Volume 1200 μL; Injection Volume 800 μL; Injection Volume 400 μL; Injection Speed at 450 μL/s; Injection Speed at 300 μL/s; Injection Speed at 150 μL/s: Backflow (uL) was assessed in the abdomen following administration of 4 different injection volumes (400, 800, 1200 and 1600 µL) at 3 different injection speeds (150, 300 and 450 µL/s), and in the thighs following administration of the selected combinations of injection volume (µL) and speed (µL/s) (400/150, 400/450, 800/300, 1600/150, 1600/450).
Arm/Group | Abdomen: Injection Region-12 s.c Injections+1 Needle Insertion | Injection Volume 1600 μL | Injection Volume 1200 μL | Injection Volume 800 μL | Injection Volume 400 μL | Injection Speed at 450 μL/s | Injection Speed at 300 μL/s | Injection Speed at 150 μL/s
Number analyzed (Participants) | 82 | 82 | 82 | 82 | 82 | 82 | 82 | 82
mcL
  Needle insertion | 0.0 (0.1) | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered
  Injection speed at 150 μL/s | NA (NA) — Not administered | 2.3 (5.1) | 0.9 (1.9) | 0.5 (1.4) | 0.6 (1.8) | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — No summary statistics done for this combination
  Injection speed at 300 μL/s | NA (NA) — Not administered | 1.4 (2.9) | 0.8 (1.9) | 0.5 (1.6) | 0.4 (1.3) | NA (NA) — Not administered | NA (NA) — No summary statistics done for this combination | NA (NA) — Not administered
  Injection speed at 450 μL/s | NA (NA) — Not administered | 0.6 (1.1) | 1.1 (4.6) | 0.5 (1.3) | 0.9 (2.7) | NA (NA) — No summary statistics done for this combination | NA (NA) — Not administered | NA (NA) — Not administered
Statistical Analysis 1: Comparison: Injection Volume 400 μL vs Injection Speed at 150 μL/s; Backflow (absorbed amount of liquid 2 minutes (±30 sec) after the injection with filter-paper rated according to the liquid scale) was analysed using a mixed ANOVA approach and calculated as the mean differences in backflow in the abdomen at different volume and speed combinations; Test type: Superiority or Other; Least Square Mean Difference = 0.6, 95% CI [-0.6 to 1.8]
Statistical Analysis 2: Comparison: Injection Volume 400 μL vs Injection Speed at 300 μL/s; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 0.4, 95% CI [-0.8 to 1.6]
Statistical Analysis 3: Comparison: Injection Volume 400 μL vs Injection Speed at 450 μL/s; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 0.9, 95% CI [-0.4 to 2.1]
Statistical Analysis 4: Comparison: Injection Volume 800 μL vs Injection Speed at 150 μL/s; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 0.5, 95% CI [-0.8 to 1.7]
Statistical Analysis 5: Comparison: Injection Volume 800 μL vs Injection Speed at 300 μL/s; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 0.5, 95% CI [-0.8 to 1.7]
Statistical Analysis 6: Comparison: Injection Volume 800 μL vs Injection Speed at 450 μL/s; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 0.5, 95% CI [-0.7 to 1.8]
Statistical Analysis 7: Comparison: Injection Volume 1200 μL vs Injection Speed at 150 μL/s; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 0.9, 95% CI [-0.3 to 2.1]
Statistical Analysis 8: Comparison: Injection Volume 1200 μL vs Injection Speed at 300 μL/s; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 0.8, 95% CI [-0.4 to 2.0]
Statistical Analysis 9: Comparison: Injection Volume 1200 μL vs Injection Speed at 450 μL/s; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 1.1, 95% CI [-0.1 to 2.3]
Statistical Analysis 10: Comparison: Injection Volume 1600 μL vs Injection Speed at 150 μL/s; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 2.3, 95% CI [1.0 to 3.5]
Statistical Analysis 11: Comparison: Injection Volume 1600 μL vs Injection Speed at 300 μL/s; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 1.4, 95% CI [0.2 to 2.6]
Statistical Analysis 12: Comparison: Injection Volume 1600 μL vs Injection Speed at 450 μL/s; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 0.6, 95% CI [-0.6 to 1.8]

6. Secondary Outcome: Estimated Mean Differences in the Volume of Backflow (uL) in the Thighs After Different Injection Volumes and Speeds as Compared to Needle Insertion
Description: as for outcome 5
Time Frame: 2 minutes (±30sec) after each injection
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcL
Groups:
- Thighs: Injection Region-5 s.c Injections+1 Needle Insertion: Backflow (uL) was assessed in each subject for the 5 s.c injections+1 needle insertion administered in the thighs.
Arm/Group | Thighs: Injection Region-5 s.c Injections+1 Needle Insertion | Injection Volume 1600 μL | Injection Volume 800 μL | Injection Volume 400 μL | Injection Speed at 450 μL/s | Injection Speed at 300 μL/s | Injection Speed at 150 μL/s
Number analyzed (Participants) | 82 | 82 | 82 | 82 | 82 | 82 | 82
mcL
  Needle insertion | 0.8 (5.6) | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Not administered
  Injection speed at 150 μL/s | NA (NA) — Not administered | 5.6 (8.6) | NA (NA) — Not administered | 1.0 (3.1) | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — No summary statistics done for this combination.
  Injection speed at 300 μL/s | NA (NA) — Not administered | NA (NA) — Not administered | 2.3 (7.9) | NA (NA) — Not administered | NA (NA) — Not administered | NA (NA) — Summary statistics is same as presented in Injection speed at 300 μL/s x Injection Volume 800 μL. | NA (NA) — Not administered
  Injection speed at 450 μL/s | NA (NA) — Not administered | 2.5 (4.6) | NA (NA) — Not administered | 1.6 (4.9) | NA (NA) — No summary statistics done for this combination. | NA (NA) — Not administered | NA (NA) — Not administered
Statistical Analysis 1: Comparison: Injection Volume 400 μL vs Injection Speed at 150 μL/s; Backflow (absorbed amount of liquid 2 minutes (±30 sec) after the injection with filter-paper rated according to the liquid scale) was analysed using a mixed ANOVA approach and calculated as the mean differences in backflow in the thigh at different volume and speed combinations; Test type: Superiority or Other; Least Square Mean Difference = 0.3, 95% CI [-0.9 to 1.5]
Statistical Analysis 2: Comparison: Injection Volume 400 μL vs Injection Speed at 450 μL/s; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 0.8, 95% CI [-0.4 to 2.1]
Statistical Analysis 3: Comparison: Injection Volume 800 μL vs Injection Speed at 300 μL/s; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 1.6, 95% CI [0.3 to 2.8]
Statistical Analysis 4: Comparison: Injection Volume 1600 μL vs Injection Speed at 150 μL/s; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 4.9, 95% CI [3.7 to 6.1]
Statistical Analysis 5: Comparison: Injection Volume 1600 μL vs Injection Speed at 450 μL/s; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 1.7, 95% CI [0.5 to 2.9]

ADVERSE EVENTS:
Time Frame: From Day 0 when receiving 19 injections and up to 48 hours after last injection.
Description: All randomised subjects receiving at least one injection (possibly needle insertion only) were included in the safety analysis set.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to defer the release of data until specified milestones are reached, for example when the clinical trial report is available. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.